CLINICAL TRIAL: NCT03788291
Title: Phase II Study of Acalabrutinib and High Frequency Low Dose Subcutaneous Rituximab in Patients With Previously Untreated CLL/SLL
Brief Title: Acalabrutinib and High Frequency Low Dose Subcutaneous Rituximab in Patients With Previously Untreated Chronic Lymphocytic Leukemia / Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Paul Barr, Director of the Clinical Trials Office for Wilmot Cancer Institute, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULYM18086
Record Dates: First submitted 2018-12-24; First posted 2018-12-27 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Phase II; Acalabrutinib; Rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acalabrutinib and Rituximab treatment (Experimental): Rituximab: administered 2 times weekly for 6 cycles. Initial dose day 1: 50 mg IV, Then 50 mg SQ thereafter.
  Acalabrutinib: 100 mg po BID starting on day 8 of cycle 1.
  * Patients who have attained a complete response who are also MRD negative at cycle 12 will undergo a BM biopsy to confirm CR and MRD negatively. If confirmed, the patient will stop therapy and be followed until disease progression.
  * Patients not in a MRD negative CR, will continue acalabrutinib.
  * Repeat response assessments (CTs, MRD testing in blood) will be performed at 24 cycles of therapy for those continuing on acalabrutinib. If both negative the patient will undergo a BM biopsy to confirm CR and MRD negativity. If confirmed, the patient will stop therapy and be followed until disease progression. In the absence of a CR or if MRD +, acalabrutinib may be continued until disease progression, unacceptable toxicity or physician/patient discretion.
  Interventions: Drug: Acalabrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — 100 mg by mouth twice a day starting on day 8 of cycle 1
Drug: Rituximab — Administered 2 times weekly for 6 cycles. Initial dose day 1: 50 mg IV, then 50 mg SQ thereafter.

SUMMARY:
The main purpose of this research study is to find out if the combination of acalabrutinib and high frequency low dose subcutaneous rituximab is safe and effective in patients who have previously untreated chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL).

DETAILED DESCRIPTION:
Despite an array of available therapies, CLL remains an incurable disease. Furthermore, the presence of certain cytogenetic abnormalities and high-risk mutational features predicts for a reduced response to treatment, and as a result, a shorter period of progression-free survival. The development of a well-tolerated more effective, easily administered and limited duration therapy would be a major contribution to the management of CLL and other B cell malignancies.

Acalabrutinib is an imidazopyrazine analogue and a potent inhibitor of BTK in vitro and in vivo. Acalabrutinib shows improved selectivity for BTK compared with ibrutinib. Functional inhibition of non-target cells (eg, T cells, NK cells, platelets) was not observed for acalabrutinib at clinically relevant concentrations. Rituximab is a chimeric monoclonal antibody targeting CD20 FDA approved for the treatment of CLL/SLL using intravenous or subcutaneous formulations.

Antibody dependent cellular phagocytosis may be optimized using high frequency subcutaneous administration of anti-CD20 monoclonal antibodies. Unlike ibrutinib, acalabrutinib does not cause significant in vitro inhibition of rituximab induced antibody dependent cellular phagocytosis in vitro. The investigator thus proposes that acalabrutinib would be an ideal partner drug with high frequency low dose SQ rituximab in the treatment of CLL and that the combination will increase the efficacy of therapy for CLL patients by decreasing the time to achievement of complete response and allowing for shorter and less toxic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of B-cell CLL or SLL, with diagnosis established according to IWCLL criteria and documented within medical records. Patients must not have received previous therapy for CLL/SLL
2. CLL/SLL that warrants treatment consistent with accepted IWCLL criteria for initiation of therapy. Any one of the following conditions constitutes CLL/SLL that warrants treatment:

   1. Evidence of progressive marrow failure as manifested by the onset or worsening of anemia and/or thrombocytopenia, or
   2. Massive (i.e., lower edge of spleen ≥6 cm below the left costal margin), progressive, or symptomatic splenomegaly, or
   3. Massive (i.e., ≥10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy, or
   4. Progressive lymphocytosis in the absence of infection, with an increase in blood absolute lymphocyte count (ALC) ≥50% over a 2-month period or lymphocyte doubling time of <6 months (as long as initial ALC was ≥30,000/L), or
   5. Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy, or
   6. Constitutional symptoms, defined as any one or more of the following disease-related symptoms or signs occurring in the absence of evidence of infection:

   i. Unintentional weight loss of ≥10% within the previous 6 months, or

   ii. Significant fatigue (≥Grade 2), or

   iii. Fevers >100.5°F or 38.0°C for ≥2 weeks, or

   iv. Drenching night sweats for >1 month.
3. Adequate organ system function, defined as follows:

   1. Absolute neutrophil count (ANC) ≥ 0.5x109/L and platelet count ≥ 30x109/L
   2. Total bilirubin ≤2.5 times the upper limit of normal (ULN) unless due to Gilbert's disease
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN if no liver involvement or ≤5 x the ULN if known liver involvement
   4. Calculated creatinine clearance >30 mL/min (as calculated by the Cockcroft-Gault formula)
   5. Patients with PT/INR or aPTT ≤2xULN.
4. ECOG performance status ≤ 2 unless related to CLL.
5. Male or female ≥ 18 years of age.
6. Ability to swallow and retain oral medication.
7. Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib and for 12 months following last dose of rituximab. (see Appendix 3 for examples)
8. Willingness and ability to comply with study and follow-up procedures, and give written informed consent.

Exclusion Criteria:

1. Patients receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery).

   a. Systemic corticosteroid therapy started prior to study entry is allowed as clinically warranted. Topical or inhaled corticosteroids are permitted.
2. Serologic status reflecting active hepatitis B or C infection. Patients who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.
3. Known history of HIV.
4. Known histological transformation from CLL to an aggressive lymphoma.
5. Evidence of ongoing systemic bacterial, fungal or viral infection, except localized fungal infections of skin or nails. NOTE: Patients may be receiving prophylactic antiviral or antibacterial therapies at investigator discretion.
6. Live virus vaccines within 4 weeks prior to C1D1 or during rituximab therapy.
7. History of anaphylaxis (excluding infusion related reactions) in association with previous anti-CD20 administration or acalabrutinib.
8. Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

   1. Symptomatic, or history of documented congestive heart failure (NY Heart Association functional classification III-IV)
   2. Uncontrolled cardiac arrhythmia (Patients with controlled atrial fibrillation/flutter are eligible)
   3. Myocardial infarction within 3 months of enrollment
   4. Angina not well-controlled by medication
   5. Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac/vascular stenting within 3 months of enrollment.
   6. Active bleeding or history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
   7. Any history of intracranial bleed or stroke within 6 months of first dose of study drug
   8. Patients with suspected or confirmed PML
   9. Patients with malabsorption syndrome or gastrointestinal disease that limits absorption of oral medication
9. Malignancy within 2 years of study enrollment except for adequately treated basal, squamous cell carcinoma or non-melanomatous skin cancer, carcinoma in situ of the cervix, superficial bladder cancer not treated with intravesical chemotherapy or BCG within 6 months, localized prostate cancer and PSA <1.0 mg/dL on 2 consecutive measurements at least 3 months apart with the most recent one being within 4 weeks of study entry.
10. Patients with active uncontrolled autoimmune hemolytic anemia or ITP.
11. Inability to discontinue use of strong CYP3A inhibitors. Patients taking moderate CYP3A inhibitors or strong CYP3A inducers are eligible.
12. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days of first dose of study drug.
13. Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole) at study entry. Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Barr, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Wallace DS, Zent CS, Baran AM, Reagan PM, Casulo C, Rice G, Friedberg JW, Barr PM. Acalabrutinib and high-frequency low-dose subcutaneous rituximab for initial therapy of chronic lymphocytic leukemia. Blood Adv. 2023 Jun 13;7(11):2496-2503. doi: 10.1182/bloodadvances.2022009382. PMID 36689726

RESULTS

PARTICIPANT FLOW:
Groups:
- Acalabrutinib and Rituximab Treatment: Rituximab: administered 2 times weekly for 6 cycles. Initial dose day 1: 50 mg IV, Then 50 mg SQ thereafter.
  Acalabrutinib: 100 mg po BID starting on day 8 of cycle 1.
  * Patients who have attained a complete response who are also MRD negative at cycle 12 will undergo a BM biopsy to confirm CR and MRD negatively. If confirmed, the patient will stop therapy and be followed until disease progression.
  * Patients not in a MRD negative CR, will continue acalabrutinib.
  * Repeat response assessments (CTs, MRD testing in blood) will be performed at 24 cycles of therapy for those continuing on acalabrutinib. If both negative the patient will undergo a BM biopsy to confirm CR and MRD negativity. If confirmed, the patient will stop therapy and be followed until disease progression. In the absence of a CR or if MRD +, acalabrutinib may be continued until disease progression, unacceptable toxicity or physician/patient discretion.
  Acalabrutinib: 100 mg by mouth twice a day starting on day 8 of cycle 1
  Rituximab: Administered 2 times weekly for 6 cycles. Initial dose day 1: 50 mg IV, then 50 mg SQ thereafter.
Period: Overall Study
Arm/Group | Acalabrutinib and Rituximab Treatment
Started | 38 (39 participants were consented, but 1 participant was found to have a non-CLL B-cell non-Hodgkin lymphoma and was excluded from all data collection.)
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acalabrutinib and Rituximab Treatment
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 66.5 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a Complete Response Rate (CR) at 1 Year of Therapy
Description: To satisfy criteria for a CR, all of the following criteria must be met:
  * No evidence of new disease
  * ALC in peripheral blood of <4 x 109/L
  * Regression of all target nodal masses to normal size ≤1.5 cm in the LD
  * Normal spleen and liver size
  * Regression to normal of all nodal non-target disease and disappearance of all detectable non-nodal, non-target disease
  * Morphologically negative bone marrow defined as <30% of nucleated cells being lymphoid cells and no lymphoid nodules in a bone marrow sample (the presence of benign reactive nodules is still compatible with a CR)
  * Absence of constitutional symptoms
  * Peripheral blood counts meeting all of the following criteria:
    * ANC >1.5 x 109/L without need for exogenous growth factors (e.g., G-CSF)
    * Platelet count ≥100 x 109/L without need for exogenous growth factors
    * Hemoglobin ≥110 g/L (11.0 g/dL) without red blood cell transfusions or need for exogenous growth factors (e.g., erythropoietin)
Time Frame: 1 year
Measure: Number; unit: proportion of participants
Arm/Group | Acalabrutinib and Rituximab Treatment
Number analyzed (Participants) | 38
proportion of participants | 0.26

2. Secondary Outcome: Proportion of Subjects With Minimal Residual Disease in Peripheral Blood and Bone
Description: 6-color flow cytometry was performed on patients achieving a complete response to evaluate for minimal residual disease.
Time Frame: 1 year
Population: This analysis was only performed on participants with a complete response after 12 cycles of treatment. Ten participants had a complete response.
Measure: Number; unit: proportion or participants
Arm/Group | Acalabrutinib and Rituximab Treatment
Number analyzed (Participants) | 10
proportion or participants | 1.0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Acalabrutinib and Rituximab Treatment
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 10/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acalabrutinib and Rituximab Treatment (N=38)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 1
COVID-19 infection (Infections and infestations) | 4
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Joint Infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Coronary artery disease (Cardiac disorders) | 1
Stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acalabrutinib and Rituximab Treatment (N=38)
Anemia (Blood and lymphatic system disorders) | 2
COVID-19 (Infections and infestations) | 15
Pneumonia (non-COVID) (Infections and infestations) | 5
Dental Infection (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 3
Upper respiratory infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 8
arthritis/arthralgias (Musculoskeletal and connective tissue disorders) | 15
bruising (Musculoskeletal and connective tissue disorders) | 15
hematoma (Musculoskeletal and connective tissue disorders) | 4
Myalgias (Musculoskeletal and connective tissue disorders) | 19
Rash (Musculoskeletal and connective tissue disorders) | 9
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 11
Cough (General disorders) | 10
Dizziness (Nervous system disorders) | 8
Edema (General disorders) | 12
Fatigue (General disorders) | 14
Headache (Nervous system disorders) | 26
Infusion reaction (Injury, poisoning and procedural complications) | 24
Injection site reaction (General disorders) | 12
Sinus bradychardia (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03788291/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03788291/ICF_001.pdf